CLINICAL TRIAL: NCT02039947
Title: BRF117277: A Phase II, Open-Label, Multicentre Study of Dabrafenib Plus Trametinib in Subjects With BRAF Mutation-Positive Melanoma That Has Metastasized to the Brain
Brief Title: Study to Evaluate Treatment of Dabrafenib Plus Trametinib in Subjects With BRAF Mutation-Positive Melanoma That Has Metastasized to the Brain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 117277
Record Dates: First submitted 2013-12-19; First posted 2014-01-20 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Melanoma and Brain Metastases
Keywords: BRAF V600K mutation; Metastatic Melanoma; BRAF V600R mutation; BRAF V600D mutation; BRAF V600E mutation; Brain metastases BRAF inhibitor; Intracranial
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Subjects will receive dabrafenib 150 milligram (mg) twice daily and trametinib 2 mg once daily until evidence of disease progression, death, or unacceptable toxicity.
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Cohort B (Experimental): Subjects will receive dabrafenib 150 mg twice daily and trametinib 2 mg once daily until evidence of disease progression, death, or unacceptable toxicity
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Cohort C (Experimental): Subjects will receive dabrafenib 150 mg twice daily and trametinib 2 mg once daily until evidence of disease progression, death, or unacceptable toxicity
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Cohort D (Experimental): Subjects will receive dabrafenib 150 mg twice daily and trametinib 2 mg once daily until evidence of disease progression, death, or unacceptable toxicity
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib will be provided as 50 mg and 75 mg capsules
Drug: Trametinib — Trametinib will be provided as 0.5 mg and 2.0 mg tablets

SUMMARY:
This is a multi-cohort, open label, Phase II study with Dabrafenib (GSK2118436) and Trametinib (GSK1120212) combination therapy in subject with BRAF mutation-positive melanoma that has metastasized to the brain. This study will evaluate the safety and efficacy of 4 cohorts. Cohorts will consist of; V600 E, D, K, R mutations, metastases to the brain, symptomatic and asymptomatic, with or without prior local (brain) therapy, with or without prior local (brain) therapy, and range of ECOG scores from 0-2.

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status range of 0-2
* Histologically confirmed cutaneous metastatic melanoma of V600 E, K, D or R.
* May be systemic naïve or received up to two previous systemic treatment regimens for metastatic melanoma.
* Must be able to undergo MRI and have at least one measurable intracranial lesion for which specific criteria have to be met.

Exclusion Criteria:

* Prior treatment with any BRAF inhibitor or any mitogen-activated protein/extracellular signal-regulated kinase inhibitor.
* Anti-cancer therapy or investigational anti-cancer therapy or chemotherapy without delayed toxicity within treatment specific timeframe.
* Treatment with stereotactic radiosurgery or treatment with whole-brain radiation within treatment specific timeframe.
* Any presence of leptomeningeal disease or any parenchymal brain metastasis
* History of another malignancy, some exceptions may apply.
* A history or evidence of cardiovascular risk- specific criteria have to be met
* A history or current evidence/risk of retinal vein occlusion or retinal pigment epithelial detachment - specific criteria have to be met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-02-21 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- United States (10):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
- Australia (3):
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Greenslopes, Queensland
  - Novartis Investigative Site, Melbourne, Victoria
- Canada (4):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (11):
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (7):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Tübingen, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Kiel, Schleswig-Holstein
  - Novartis Investigative Site, Gera, Thuringia
- Italy (2):
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Padua, Veneto
- Spain (8):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza

REFERENCES:
- [Derived] Syeda MM, Wiggins JM, Corless BC, Long GV, Flaherty KT, Schadendorf D, Nathan PD, Robert C, Ribas A, Davies MA, Grob JJ, Gasal E, Squires M, Marker M, Garrett J, Brase JC, Polsky D. Circulating tumour DNA in patients with advanced melanoma treated with dabrafenib or dabrafenib plus trametinib: a clinical validation study. Lancet Oncol. 2021 Mar;22(3):370-380. doi: 10.1016/S1470-2045(20)30726-9. Epub 2021 Feb 12. PMID 33587894
- [Derived] Davies MA, Saiag P, Robert C, Grob JJ, Flaherty KT, Arance A, Chiarion-Sileni V, Thomas L, Lesimple T, Mortier L, Moschos SJ, Hogg D, Marquez-Rodas I, Del Vecchio M, Lebbe C, Meyer N, Zhang Y, Huang Y, Mookerjee B, Long GV. Dabrafenib plus trametinib in patients with BRAFV600-mutant melanoma brain metastases (COMBI-MB): a multicentre, multicohort, open-label, phase 2 trial. Lancet Oncol. 2017 Jul;18(7):863-873. doi: 10.1016/S1470-2045(17)30429-1. Epub 2017 Jun 4. PMID 28592387

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A subject was considered to have completed the study if the subject died during the study treatment or follow-up period or (for subject in Cohort A) had at least 3 years follow-up from the date of first dose of study treatment at the end of the study.
  All subjects achieved that definition and then the study ended.
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D
Started | 76 | 16 | 16 | 17
Completed | 76 | 16 | 16 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Total
Number analyzed (Participants) | 76 | 16 | 16 | 17 | 125
Age, Continuous [Median (Standard Deviation); unit: Years] | 53.2 (14.69) | 55.1 (11.05) | 65.6 (10.40) | 47.5 (13.01) | 54.2 (14.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 6 | 5 | 6 | 53
  Male | 40 | 10 | 11 | 11 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 76 | 16 | 16 | 17 | 125
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Response (IR) Rate in Cohort A
Description: The intracranial response rate is defined as the percentage of subjects achieving a confirmed intracranial CR or PR. This is based on investigator-assessed best intracranial response.
Time Frame: From the start of treatment until disease progression or the start of new anti-cancer therapy
Population: All Treated population - All subjects who receive at least one dose of study medication are comprised the All Treated subjects (ATS) population.
Measure: Number; unit: Number of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 76
Number of participants | 45
Statistical Analysis 1: Comparison: Cohort A; Test type: Superiority; p < .0001, percent; Response rate = 59, 95% CI 2-sided [47.3 to 70.4] — Percent

2. Secondary Outcome: Intracranial Response Rate of Cohorts B, C and D
Description: The intracranial response rate is defined as the percentage of subjects achieving a confirmed intracranial CR or PR. This is based on investigator-assessed best intracranial response. No hypothesis testing completed for cohort A, B,C and D
Time Frame: Approximately 2 years
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Cohort B | Cohort C | Cohort D
Number analyzed (Participants) | 16 | 16 | 17
Number of participants | 9 | 7 | 10

3. Secondary Outcome: Disease Control for Intracranial, Extracranial and Overall Response for Each Cohort
Description: Disease Control rate is defined as the percentage of subjects achieving a confirmed intracranial/extracranial/overall CR or PR or SD or Non-CR/Non-PD. This is based on investigator-assessed response. No hypothesis testing completed for cohort A, B,C and D
Time Frame: Approximately 2 years
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D
Number analyzed (Participants) | 76 | 16 | 16 | 17
Number of participants
  Intracranial | 59 | 14 | 12 | 15
  Extra cranial | 60 | 11 | 15 | 11
  Overall rate | 60 | 14 | 12 | 15

4. Secondary Outcome: Extracranial Response Rate (ER) for Each Cohort
Description: Extracranial Response Rate was defined as the percentage of participants with Complete response (CR) or Partial response (PR) at anytime. This is based on investigator-assessed response. No hypothesis testing completed for cohort A,B,C and D
Time Frame: Approximately 2 years
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D
Number analyzed (Participants) | 76 | 16 | 16 | 17
Number of participants | 42 | 7 | 12 | 7

5. Secondary Outcome: Overall Response (OR) for Each Cohort
Description: the number of subjects with a confirmed overall Complete response (CR) or Partial response (PR) by investigator assessment using the Response evaluation criteria in solid tumors (RECIST 1.1 criteria). To determine the overall response, all target and non-target lesions will be assessed using modified RECIST 1.1 criteria.
Time Frame: Approximately 2 years
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D
Number analyzed (Participants) | 76 | 16 | 16 | 17
Number of participants | 45 | 9 | 7 | 11

6. Secondary Outcome: Duration of Intracranial, Extracranial and Overall Response for Each Cohort
Description: Duration of intracranial, extracranial and overall response, are defined as the time from first documented evidence of CR or PR until time of first documented intracranial, extracranial, or overall disease progression. No hypothesis testing completed for cohort A,B,C and D
Time Frame: From first documented evidence of CR or PR until time of first documented intracranial, extracranial, or overall disease progression
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D
Number analyzed (Participants) | 76 | 16 | 16 | 17
Month
  Duration of intracranial | 6.5 [4.9 to 8.6] | 7.3 [3.6 to 12.6] | 8.3 [1.3 to 15.0] | 4.5 [2.8 to 5.9]
  Duration of extracranial | 10.2 [5.8 to NA] — Upper Limit not reachable. | NA [NA to NA] — Lower and upper Limit not reachable. | 4.9 [3.0 to 22.4] | 5.9 [1.8 to NA] — Upper Limit not reachable.
  Duration of Overall Response | 6.2 [4.9 to 8.3] | 12.5 [5.3 to NA] — Upper Limit not reachable. | 6.6 [1.3 to 16.3] | 4.5 [2.8 to 11.2]

7. Secondary Outcome: Progression-free Survival (PFS) for Each Cohort Based on Investigator Assessment
Description: PFS is defined as the interval between first dose and the earliest date of disease progression or death due to any cause. No hypothesis testing completed for cohort A,B,C and D
Time Frame: From the first dose to the earliest date of disease progression or death
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D
Number analyzed (Participants) | 76 | 16 | 16 | 17
Month | 5.7 [5.3 to 7.3] | 7.2 [4.7 to 14.6] | 3.7 [1.7 to 6.5] | 5.5 [3.7 to 11.6]

8. Secondary Outcome: Overall Survival (OS) for Each Cohort
Description: Overall survival (OS) is defined as the time from the first dose until death due to any cause. No hypothesis testing completed for cohort A,B,C and D
Time Frame: From the first dose to death
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D
Number analyzed (Participants) | 76 | 16 | 16 | 17
Month | 10.8 [8.7 to 17.9] | 24.3 [7.9 to NA] — NA - Not reachable | 10.1 [4.6 to 17.6] | 11.5 [6.8 to 22.4]

ADVERSE EVENTS:
Time Frame: every 12 weeks until death up to 4 years
Description: AE additional description
Groups:
- Total: Total
Arm/Group | Cohort A | Cohort B | Cohort C | Cohort D | Total
All-Cause Mortality (participants affected / at risk) | 54/76 | 10/16 | 15/16 | 13/17 | 92/125
Serious Adverse Events (participants affected / at risk) | 26/76 | 5/16 | 4/16 | 9/17 | 44/125
Other Adverse Events (participants affected / at risk) | 74/76 | 16/16 | 16/16 | 17/17 | 123/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=76) | Cohort B (N=16) | Cohort C (N=16) | Cohort D (N=17) | Total (N=125)
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Detachment of retinal pigment epithelium (Eye disorders) | 1 | 0 | 0 | 0 | 1
Macular detachment (Eye disorders) | 1 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 1 | 0 | 2
Malaise (General disorders) | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 1 | 2 | 2 | 9
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 2 | 0 | 1 | 2 | 5
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 1
Troponin T increased (Investigations) | 1 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 2
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 2 | 0 | 0 | 1 | 3
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=76) | Cohort B (N=16) | Cohort C (N=16) | Cohort D (N=17) | Total (N=125)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 2 | 6
Lymphopenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 11 | 2 | 1 | 0 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 1 | 2 | 7
Cyanosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 1 | 0 | 4
Asthenopia (Eye disorders) | 0 | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 1
Conjunctival irritation (Eye disorders) | 0 | 0 | 0 | 1 | 1
Diplopia (Eye disorders) | 1 | 0 | 1 | 1 | 3
Dry eye (Eye disorders) | 2 | 0 | 0 | 1 | 3
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 2 | 3
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 0 | 2
Posterior capsule opacification (Eye disorders) | 0 | 0 | 1 | 0 | 1
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 1 | 1
Retinopathy (Eye disorders) | 0 | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 3 | 1 | 1 | 1 | 6
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0 | 2 | 3
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 1 | 1
Vitreous floaters (Eye disorders) | 3 | 1 | 0 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 1 | 0 | 5 | 14
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 0 | 1 | 7
Constipation (Gastrointestinal disorders) | 8 | 1 | 4 | 6 | 19
Diarrhoea (Gastrointestinal disorders) | 24 | 8 | 3 | 7 | 42
Dry mouth (Gastrointestinal disorders) | 5 | 2 | 1 | 3 | 11
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 1 | 0 | 8
Faecalith (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3
Nausea (Gastrointestinal disorders) | 24 | 7 | 4 | 6 | 41
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 4
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 6
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 24 | 2 | 2 | 6 | 34
Asthenia (General disorders) | 28 | 5 | 3 | 5 | 41
Chest pain (General disorders) | 3 | 0 | 1 | 0 | 4
Chills (General disorders) | 18 | 6 | 7 | 6 | 37
Face oedema (General disorders) | 2 | 0 | 0 | 1 | 3
Fatigue (General disorders) | 7 | 4 | 8 | 3 | 22
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 1
General physical health deterioration (General disorders) | 2 | 1 | 0 | 0 | 3
Ill-defined disorder (General disorders) | 0 | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 5 | 2 | 1 | 0 | 8
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 11 | 2 | 2 | 3 | 18
Pain (General disorders) | 2 | 1 | 0 | 1 | 4
Pyrexia (General disorders) | 45 | 7 | 8 | 8 | 68
Temperature regulation disorder (General disorders) | 1 | 1 | 0 | 0 | 2
Thirst (General disorders) | 0 | 0 | 1 | 0 | 1
Xerosis (General disorders) | 3 | 0 | 0 | 1 | 4
Hepatocellular injury (Hepatobiliary disorders) | 2 | 2 | 0 | 0 | 4
Angular cheilitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 4 | 0 | 0 | 1 | 5
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 4 | 2 | 0 | 4 | 10
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Influenza (Infections and infestations) | 7 | 0 | 0 | 0 | 7
Laryngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 2 | 0 | 0 | 1 | 3
Nasopharyngitis (Infections and infestations) | 7 | 2 | 2 | 0 | 11
Onychomycosis (Infections and infestations) | 2 | 0 | 1 | 1 | 4
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 2
Oral herpes (Infections and infestations) | 3 | 1 | 0 | 0 | 4
Paronychia (Infections and infestations) | 1 | 0 | 1 | 0 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Pulpitis dental (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Rhinitis (Infections and infestations) | 4 | 0 | 2 | 0 | 6
Sialoadenitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 2 | 1 | 0 | 0 | 3
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 | 2 | 6
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 9 | 2 | 1 | 3 | 15
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 12 | 3 | 2 | 3 | 20
Blood alkaline phosphatase increased (Investigations) | 6 | 1 | 2 | 3 | 12
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 7 | 3 | 0 | 0 | 10
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 6 | 1 | 1 | 0 | 8
Blood phosphorus decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood pressure increased (Investigations) | 1 | 1 | 0 | 0 | 2
Blood sodium increased (Investigations) | 0 | 0 | 0 | 1 | 1
C-reactive protein increased (Investigations) | 4 | 1 | 0 | 0 | 5
Ejection fraction decreased (Investigations) | 4 | 1 | 1 | 1 | 7
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 7 | 1 | 1 | 4 | 13
Lipase increased (Investigations) | 3 | 0 | 0 | 1 | 4
Neutrophil count decreased (Investigations) | 4 | 0 | 1 | 1 | 6
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 2 | 0 | 1 | 0 | 3
Weight decreased (Investigations) | 4 | 2 | 3 | 3 | 12
Weight increased (Investigations) | 4 | 0 | 0 | 2 | 6
White blood cell count decreased (Investigations) | 2 | 0 | 1 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 9 | 4 | 7 | 3 | 23
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 2 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 3 | 2 | 6 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 1 | 3 | 2 | 17
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 0 | 4 | 1 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 3 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 1 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 5 | 2 | 6 | 26
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 1 | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 3 | 3 | 2 | 16
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0 | 3
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 2
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 3
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 2
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 3 | 4
Aphonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 5 | 0 | 3 | 13
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 2 | 1 | 1 | 0 | 4
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 28 | 5 | 6 | 8 | 47
Hemianopia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 5 | 1 | 0 | 2 | 8
Paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 2 | 0 | 0 | 2
Seizure (Nervous system disorders) | 2 | 1 | 3 | 3 | 9
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Temporal lobe epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Tongue paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Tonic clonic movements (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 3 | 0 | 1 | 0 | 4
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 1 | 4
Apathy (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 1 | 3
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 1 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 6 | 0 | 0 | 2 | 8
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 3
Nocturia (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 2
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 1 | 3 | 16
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 1 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 2 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 5 | 0 | 1 | 0 | 6
Actinic elastosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 0 | 1 | 2 | 10
Aquagenic wrinkling of palms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 1 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 2 | 3 | 3 | 15
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0 | 4 | 1 | 10
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 1 | 6
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 7 | 1 | 0 | 0 | 8
Intertrigo (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1 | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 4
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0 | 4
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 2 | 9
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 9 | 7 | 3 | 3 | 22
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Skin hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 3
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 2
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 1 | 0 | 2 | 0 | 3
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 2
Hypertension (Vascular disorders) | 6 | 3 | 3 | 0 | 12
Hypotension (Vascular disorders) | 1 | 2 | 0 | 1 | 4
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 1 | 2
Peripheral venous disease (Vascular disorders) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT02039947/SAP_000.pdf
  • Study Protocol (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT02039947/Prot_001.pdf